CLINICAL TRIAL: NCT05336071
Title: Study on Bioavailability Study of INS068 Injection by Subcutaneous Injection of New and Old Formulations in Healthy Subjects
Brief Title: The Relative Bioavailability of INS068 Injection With Two Different Formulations in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: INS068-104
Record Dates: First submitted 2022-04-08; First posted 2022-04-20 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: The study is a single-centre, randomized, open, 2-period, 2-sequence crossover design clinical trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental): T - R(T: new formulation, R: old formulation)
  Interventions: Drug: INS068 injection
- Treatment group B (Experimental): R -T(T: new formulation, R: old formulation)
  Interventions: Drug: INS068 injection

INTERVENTIONS:
Drug: INS068 injection — Group A subjects were injected formulation T and formulation R of INS068 injection at Day1 and Day8.
  Arms: Treatment group A
Drug: INS068 injection — Group B subjects were injected formulation R and formulation T of INS068 injection at Day1 and Day8.
  Arms: Treatment group B

SUMMARY:
The study is a single-centre, randomized, open, 2-period, 2-sequence crossover design clinical trial. It is planned to enroll 24 healthy male subjects. Subjects will receive INS068 injection on Day1 and Day8.

ELIGIBILITY:
Inclusion Criteria:

1. The subject can communicate well with the researcher, understand and comply with the requirements of this study, and understand and sign the informed consent.
2. Healthy subjects aged 18 ~ 55 (including the boundary value), healthy male.
3. Body mass index (BMI) within the range of 18 ~ 27 kg/m2 (including the boundary value) (BMI= weight (kg)/height 2 (m2)).
4. The physical examination, vital signs, laboratory examination, 12-lead electrocardiogram, abdominal B-ultrasound, and chest radiograph are normal or have no clinical significance.

Exclusion Criteria:

1. Presence of any abnormal and clinically significant laboratory tests (blood routine, blood biochemistry, urine routine, coagulation function), Hemoglobin < 120g/L; White blood cells < 3.0 ×109/L; Platelets < 100 × 109/L;Serum creatinine > upper limit of normal (ULN);Transaminases (ALT, AST) > 2 times the upper limit of normal (2 × ULN);Alkaline phosphatase > 2 times the upper limit of normal (2 × ULN); Total bilirubin > 1.5 times the upper limit of normal (1.5× ULN) ;Fasting blood glucose >6.1mmol/L or <3.9mmol/L; HbA1c≥6.5%.

2、12-lead electrocardiogram (ECG) showed abnormal and clinically significant. 3、Hepatitis B surface antigen positive, hepatitis C antibody positive. 4、Positive human immunodeficiency virus (HIV) serology and positive syphilis serology.

5、Have a history of hypertension, or have a systolic blood pressure of 90-139 mmHg or a diastolic blood pressure outside the range of 60-89 mmHg at screening.

6、Life-threatening disease (cancer other than basal cell skin cancer or squamous cell skin cancer) within 5 years.

7、Severe infectious disease of vital organs within 1 month before screening. 8、History of serious cardiovascular disease, including decompensated heart failure (NYHA class III and IV), unstable angina, stroke or transient ischemic attack, myocardial infarction, persistent and clinically significant rhythm Abnormal, or have undergone coronary artery bypass grafting or percutaneous coronary intervention, etc..

9、Use of prescription drugs (topical eye/nasal drops and creams and occasional antipyretic and analgesic drugs such as acetaminophen within recommended doses are permitted) and over-the-counter drugs, dietary supplements, vitamins, and Chinese herbal medicine (regular vitamins are allowed).

10、A history of recurrent or severe drug food allergy, or known or suspected allergy to any component of the study drug.

11、Those who have participated in any drug clinical trials within 3 months before screening, who participated in clinical trials are defined as: those who have used test drugs; The elder shall prevail).

12、Alcoholism within 3 months prior to screening (average ≥14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine); alcohol or alcohol consumption within 48 hours prior to dosing Gas test result is positive.

13、Smokers (at least 5 cigarettes per day in the 1 year prior to screening) or non-smokers (less than 5 cigarettes per day in the 1 year prior to screening) who smoked (including nicotine replacement use) within 48 hours prior to dosing; during the trial Inability or unwillingness to smoke, nicotine gum, or transdermal nicotine patches.

14、Drinking/eating coffee, tea, chocolate or soft drinks such as cola containing methylxanthines (theophylline, caffeine or theobromine) long-term or within 48 hours before administration.

15、Do vigorous exercise, such as weightlifting, sprinting, long-distance running, cycling, swimming, football, etc., within 48 hours before administration.

16、Known or suspected history of drug abuse or positive urine drug screening test within 5 years prior to screening.

17、Donate blood within 1 month before screening; or donate blood ≥ 400 mL within 3 months before screening, or have trauma or major surgical operation with blood loss ≥ 400 mL.

18、Mentally incapacitated or language-impaired subjects who cannot adequately understand or participate in the trial process.

19、The investigator evaluates that the subject has poor compliance or the condition of the vein in the arm cannot draw blood, or has a history of fainting blood and needles.

20、Males of childbearing potential but unwilling to use contraception during the trial and for four weeks after administration.

21、At the discretion of the investigator, there are any other circumstances that interfere with the conduct of the trial or the assessment of the results.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2022-05-26 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
Maximum observed serum concentration (Cmax) of INS068 injection | from Day1 to Day5 after the first cycle（each cycle is 5 days） and from Day8 to Day12 after the second cycle（each cycle is 5 days）
Area under the plasma concentration versus time curve (AUC0-t) of INS068 injection | from Day1 to Day5 after the first cycle（each cycle is 5 days） and from Day8 to Day12 after the second cycle（each cycle is 5 days）
Area under the plasma concentration versus time curve (AUC0-inf ) of INS068 injection | from Day1 to Day5 after the first cycle（each cycle is 5 days） and from Day8 to Day12 after the second cycle（each cycle is 5 days）

SECONDARY OUTCOMES:
Time to maximum observed serum concentration (Tmax) of INS068 injection | from Day1 to Day5 after the first cycle（each cycle is 5 days） and from Day8 to Day12 after the second cycle（each cycle is 5 days）
Time to elimination half-life (T1/2) of INS068 injection | from Day1 to Day5 after the first cycle（each cycle is 5 days） and from Day8 to Day12 after the second cycle（each cycle is 5 days）
The Clearance (CL/F) of INS068 injection | from Day1 to Day5 after the first cycle（each cycle is 5 days） and from Day8 to Day12 after the second cycle（each cycle is 5 days）
The apparent volume of distribution (Vz/F) of INS068 injection | from Day1 to Day5 after the first cycle（each cycle is 5 days） and from Day8 to Day12 after the second cycle（each cycle is 5 days）
Number of subjects with adverse events and the severity of adverse events | from Day1 to Day16 after the first dose

CONTACTS AND LOCATIONS:
Locations (1):
- The Qian Foshan Hospital of Shandong Province, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen KG, Zhang YH, Ye PP, Gao XH, Song LL, Zhou HY, Li Q, Zhao FR, Shi JY, Yang XM, Shen K, Feng S, Zhao W. Pharmacokinetics and bioavailability of a new long-acting insulin analog in healthy Chinese volunteers: an open, randomized, single-dose, two-period and two-sequence cross-over study. Front Pharmacol. 2023 Dec 22;14:1294810. doi: 10.3389/fphar.2023.1294810. eCollection 2023. PMID 38186641